CLINICAL TRIAL: NCT04087083
Title: Assistive Robotic in the Elderly: Innovative Models in the Rehabilitation of the Elderly With Stroke Through Technological Innovation
Brief Title: Innovative Models in the Rehabilitation of the Elderly With Stroke Through Technological Innovation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INRCA-01-2019
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Aging Problems; Innovative Rehabilitation Treatment Based on Robotics
Keywords: stroke; robotic rehabilitation; frail elderly; gait performance; balance; risk of falling; quality of life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- technological intervention arm (Experimental): Twenty technological treatment sessions divided into 3 training sessions per week for 7 weeks.
  Interventions: Other: Technological intervention arm
- Control arm (Active Comparator): Twenty traditional treatment sessions divided into 3 training sessions per week for 7 weeks.
  Interventions: Other: Control arm

INTERVENTIONS:
Other: Technological intervention arm — Each session will include 30 minutes of traditional physical rehabilitation therapy followed by 20 minutes of robotic training (G-EO system, Reha Technology, Switzerland), an end-effector technology that simulates floor walking and stairs climbing (up and down)
  Arms: technological intervention arm
Other: Control arm — Each session will include 50 minutes of traditional physical rehabilitation therapy
  Arms: Control arm

SUMMARY:
The final goal of the present study is to propose a new approach and an innovative therapeutic plan in the post-stroke rehabilitation of elderly patients, focused on the use of robotic device, in order to obtain the beneficial effects of this treatment.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability, injury, and death in elderly people and represents a major public health problem with substantial medical and economic consequences. The incidence of stroke rapidly increases with age, doubling for each decade after age 55 years. Gait impairment is one of the most important problems after stroke and improve walking function is often a key component of any rehabilitation program. To achieve this goal, robotic gait trainer seems to be promising. In fact, some studies underline the efficacy of robotic gait training based on end-effector technology, for different diseases, in particular in stroke patients. In this randomized controlled trial, we verify the efficacy of the robotic treatment in terms of improving the gait and reducing the risk of falling and its long-term effects.

In this single blind randomized controlled trial the investigators will include 150 elderly subacute stroke patients divided in two groups to receive a traditional rehabilitation program or a robotic rehabilitation using G-EO system, an end-effector device for the gait rehabilitation, in addition to the traditional therapy. A 20 treatment sessions will be conducted, divided into 3 training sessions per week, for 7 weeks. The control group will perform traditional therapy sessions lasting 50 minutes. The technological intervention group, using G-EO system, will carry out 30 minutes of traditional therapy and 20 minutes of treatment with a robotic system. The primary outcome of the study is the evaluation of the falling risk. Secondary outcomes are the assessment of the gait improvements and the fear of falling. Further evaluations, such as length and asymmetry of the step, walking and functional status, acceptance of the technology, will be carried.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent
* Ischemic or hemorrhagic stroke within 3 months to the recruitment, proven by computerized axial tomography or nuclear magnetic resonance
* Functional Ambulation Category (FAC) score ≤ 2
* Ranking scale score ≤ 3
* Complete communication and comprehension skills, assessed during the objective examination
* Ability to stand upright, supported or unsupported, for 1 minute

Exclusion Criteria:

* Concomitant participation in other studies
* Severe hypertonus of the hip, knee, ankle of the paretic leg with a modified Ashworth scale score ≥3
* Severe hip, knee or ankle contracture or orthopedic problem affecting ambulation that would preclude passive range of motion of the paretic leg
* Deep vein thrombosis of the lower limbs
* Other cognitive, motor and sensory deficits that negatively condition robotic training
* Treatment of spasticity of the lower limb within 3 months to the start of the study or during the study
* Lack of written informed consent
* Clinical dementia rating (CDR) score ≥ 3
* Severe systemic diseases with life expectancy < 1 year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
difference in falling risk between experimental arm and control arm | before treatment, at the end of rehabilitation sessions and 6 months, 12 months and 24 months after intervention
  falling risk will be evaluated by the Tinetti performance oriented mobility assessment (POMA). Balance section of Tinetti Performance Oriented Mobility Assessment (Tinetti Performance Oriented Mobility Assessment has two subscales, Balance and Gait section.) Balance section has 9 items. Each item can be scored in a 3 point ordinal scale (0-2). "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 16. Total score is obtained by adding the individual scores.

SECONDARY OUTCOMES:
difference in gait performance between experimental arm and control arm | before treatment, at the end of rehabilitation sessions and 6 months, 12 months and 24 months after intervention
  gait performance will be evaluated by the walking speed evaluated by instrumental gait analysis
difference in fear of falling between experimental arm and control arm | before treatment, at the end of rehabilitation sessions and 6 months, 12 months and 24 months after intervention
  fear of falling will be evaluated by the Falls Efficacy Scale - International (FES-I). Higher scores represent greater the fear of falling (ranging from 16 to 64)
difference in quality of life between experimental arm and control arm: SF-12 health survey | before treatment, at the end of rehabilitation sessions and 6 months, 12 months and 24 months after intervention
  Quality of life will be measured using the Hausa SF-12 Health Survey (SF-12-H). The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS INRCA Hospital, Ancona
  - IRCCS INRCA Hospital, Fermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maranesi E, Bevilacqua R, Di Rosa M, Pelliccioni G, Di Donna V, Luzi R, Morettini M, Sbrollini A, Casoni E, Rinaldi N, Baldoni R, Lattanzio F, Burattini L, Riccardi GR. An innovative training based on robotics for older people with subacute stroke: study protocol for a randomized controlled trial. Trials. 2021 Jun 14;22(1):400. doi: 10.1186/s13063-021-05357-8. PMID 34127032